CLINICAL TRIAL: NCT05899361
Title: A Pilot Study of a Novel Imaging Protocol in Use to Identify Lymph Nodes and Organs of Interest for Surgical Dissection Within Urologic Regions of Interest.
Brief Title: A Novel Imaging Protocol in Use to Identify Lymph Nodes and Organs of Interest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Matthew Mossanen, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-668
Record Dates: First submitted 2023-03-08; First posted 2023-06-12 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Urologic Cancer; Urologic Neoplasms; Bladder Cancer; Prostate Cancer; Testicular Cancer; Kidney Cancer; Urethral Cancer; Penile Cancer
Keywords: Lymph Node Dissection; Urologic Cancer; Urologic Neoplasms; Bladder Cancer; Prostate Cancer; Testicular Cancer; Kidney Cancer; Urethral Cancer; Penile Cancer
MeSH Terms: conditions — Urologic Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Testicular Neoplasms; Kidney Neoplasms; Urethral Neoplasms; Penile Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Electromagnetic Guided Laparoscopy + Ultrasound (Experimental): This trial will investigate the use of the novel imaging protocol patients who have a confirmed cancer diagnosis in any of the following urologic regions or organs: Bladder, Prostate, Testicle, Ureter, Kidney, Urethra, Penis, and Scrotum.
  - This research study involves the use of a standard of care laparoscope and ultrasound probe. The laparoscope and ultrasound probe will have an electromagnetic sensor attached which will assist in the tracking of lymph nodes of interest or organs of interest. It is expected that the entire time to record the data will be less than 10 minutes. standard of care laparoscope and ultrasound probe
  Interventions: Device: Electromagnetic Guided Laparoscopy; Device: Ultrasound

INTERVENTIONS:
Device: Electromagnetic Guided Laparoscopy — Standard Care
Device: Ultrasound — Standard Care

SUMMARY:
This research study is a pilot clinical trial, which hypothesizes that the combination of electromagnetic tracking in conjunction with laparoscope imaging and ultrasound probe imaging will aid in reducing the complexity of both laparoscopic lymphadenectomy and/or organ removal in patients with a confirmed diagnosis of cancer in urologic regions of interest (Bladder, Prostate, Testicular, Kidney, Urethral, and Penis), by resulting in better visualization and more accurate localization of certain areas in the diseased organ or the diseased lymph node, and allowing for improved surgical and patient outcomes, fewer complications and better clinician performance.

DETAILED DESCRIPTION:
Participants in this research study, may or may not have a tumor within a urologic region of interest such as the bladder, prostate, testicle, kidney, urethra, and penis which may or may not have spread to a lymph node and have been scheduled to undergo a lymph node dissection procedure and/or organ removal surgery within one of the previously mentioned urologic regions of interest concerning for urologic cancer.

This research study involves the use of a standard of care laparoscope and ultrasound probe. The laparoscope and ultrasound probe will have an electromagnetic sensor attached which will assist in the tracking of lymph nodes of interest or organs of interest.

It is expected that the entire time to record the data will be less than 10 minutes.

A total of 10 people will take part in this research study

This study is supported by Siemens Medical USA.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before any trial-related procedure is undertaken that is not part of the standard patient management
* Subjects aged ≥ 18 years. Selected patients must have a confirmed or suspected diagnosis of disease in urologic regions of interest, with scheduled confirmatory surgical biopsy.
* Subjects must have had either of the following scans: CT, PET or MR of acceptable quality at Brigham and Women's Hospital within the past year.
* Subjects must also be scheduled to undergo lymph node dissection for a urologic cancer or organ removal of any of the following urologic regions of interest: Bladder, Prostate, Testicle, Ureter, Kidney, Urethra, Penis, and Scrotum
* Subjects must also be scheduled to undergo a laparoscopic lymph node dissection and/or a urologic organ removal within any OR at BWH.

Exclusion Criteria:

* Severely impaired renal function with an EGFR < 30 mL/min/body surface area
* Evidence of any significant, uncontrolled comorbid condition that could affect compliance with the protocol or interpretation of the results, which is to be judged at the discretion of the PI
* History of hypersensitivity or other contraindication to contrast media
* Contraindication to general anesthesia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-08-26 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Laparoscope Images | 1 year
  Laparoscope images are images recorded by the laparoscope surgical device.
Ultrasound Images | 1 year
  Ultrasound Images are images taken by an ultrasound probe.
Electromagnetic Tracking Data | 1 year
  Electromagnetic tracking data is gathered from the movements made by the laparoscope surgical device during surgery. First-order statistics measures will be computed, which include Kinematics metrics such as laparoscope path length, velocity, acceleration, and jerk.
  We will analyze the data using a mixed model regression analysis with kinematics metrics as the response and subject as the random effect. Since the kinematics measures are time series, we will address the temporal correlation in this regression model. The fixed effects in this model will include target tissue type, CT Hansfield units, surgeon assessment of navigation difficulty, and patient's BMI. We will test for kinematics outliers by applying the Grubb's test. If there are kinematics outliers, we will try to explain them by going back to the scan and patient history.

SECONDARY OUTCOMES:
Retrospective navigation accuracy | 1 year
  We are collecting data for future assessment of navigation systems, in those studies the primary out will be navigation accuracy
  We will analyze the data using a mixed model regression analysis with navigation accuracy as the response and subject as the random effect, as above. We will test for accuracy outliers by applying the Grubb's test and investigate accuracy outliers.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mossanen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation